CLINICAL TRIAL: NCT04277117
Title: Meals for Me: Drop Shipment Versus Personally Delivered Medically Tailored Meals for Patients With Unmanaged Diabetes.
Brief Title: Meals for Me: Drop Shipment Versus Personally-delivered Meals for Diabetes Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Meals on Wheels Central Texas (Other)
Responsible Party: Principal Investigator, Maninder Kahlon, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00002808-2022
Record Dates: First submitted 2020-01-31; First posted 2020-02-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: Food as Medicine; Medically tailored meals; Chronic Disease; Food Insecurity; Food Home Delivery; Implementation Science
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: Community-based trial randomized on a 2:3:3 ratio
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research staff responsible for data collection at the sites are blinded to the arm allocation of the participant. At follow-up time points, however, a set of questions is asked that are different for each of the three arms on food intake and preferences, and for arm 2, for the experience of delivery. To minimize influence of unblinding, we will actively cross-assign research staff to different locations for follow-up visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waitlisted control (Other): Phase 1 (6 months, months 1-6):
  * Educational materials on healthy eating for diabetes
  * No meal delivery
  Phase 2 (6 months, months 7-12): Standard MOWCTX home meal delivery: 5 meals a week, delivered daily 2 to 4X a week
  Interventions: Behavioral: Waitlist; Behavioral: Medically tailored meals - Standard MOWCTX delivery with human interaction
- "Daily Warm" MTM in-person delivery (Experimental): Phase 1 (6 months, months 1-6):
  * Educational materials on healthy eating for diabetes
  * 10 medically-tailored meals (MTM) per week, delivered 3-5x per week Mon-Fri
  * Each delivery day, 1 hot and 1 frozen + snack delivered to the participant's home by trained volunteers and/or paid delivery drivers who provide human interaction. Depending on the participant's availability (3-5 days/week), more frozen meals will be given one day to account for a total of 10 meals every week.
  Phase 2 (6 months, months 7-12): Standard MOWCTX home meal delivery: 5 meals a week, delivered daily 2 to 4X a week
  Interventions: Behavioral: Medically tailored meals - Daily delivery with human interaction; Behavioral: Medically tailored meals - Standard MOWCTX delivery with human interaction
- "Weekly Frozen" MTM drop shipment (Experimental): Phase 1 (6 months, months 1-6):
  * Educational materials on healthy eating for diabetes
  * 10 medically-tailored meals (MTM) delivered once a week
  * Each week all meals are frozen.
  * Meals are shipped to the participant's home with no human interaction
  Phase 2 (6 months, months 7-12): Standard MOWCTX home meal delivery: 5 meals a week, delivered daily 2 to 4X a week.
  Interventions: Behavioral: Medically tailored meals - Weekly delivery with no human interaction; Behavioral: Medically tailored meals - Standard MOWCTX delivery with human interaction

INTERVENTIONS:
Behavioral: Waitlist — Phase 1 (6 months)
  • Educational materials on such topics as healthy eating for diabetes.
  Arms: Waitlisted control
Behavioral: Medically tailored meals - Daily delivery with human interaction — Phase 1 (6 months)
  * Educational materials on such topics as healthy eating for diabetes, in addition to materials on meal planning and instructions.
  * Food: 10 MTM a week: mix of hot and frozen, and 5-10 snacks per week. Meals and snacks offer approx. 1200 kcal per day.
  * Delivery: 3 to 5x per week. Each delivery day, one meal is warm, the other is frozen. Depending on the participant's availability (3-5 days/week), more frozen meals will be given one day to account for a total of 10 meals every week.
  * Engagement: MOWCTX's trained volunteers and/or paid delivery drivers delivering the meals will have a brief social interaction (at minimum in-person hand-off & visual check) with the participant.
  Arms: "Daily Warm" MTM in-person delivery
Behavioral: Medically tailored meals - Weekly delivery with no human interaction — Phase 1 (6 months)
  * Educational materials on such topics as healthy eating for diabetes, in addition to materials on meal planning and instructions.
  * Food: 10 frozen MTM and 5-10 healthy snacks (with the goal of providing 2 meals and 1-2 snacks for 5 days of the week). Meals and snacks offer approx. 1200 kcal per day. Nutritionally similar and frequently the same meal as that delivered in the daily delivery arm.
  * Delivery: 1x per week shipment.
  * Engagement: Meals are shipped to the participant's home. No human engagement.
  Arms: "Weekly Frozen" MTM drop shipment
Behavioral: Medically tailored meals - Standard MOWCTX delivery with human interaction — Phase 2 (6 months)
  * Food: 5 MTM a week plus snacks. Planned to offer approx. 600 kcal per day.
  * Delivery: 2 to 4x a week (depending on participant availability), including daily delivery of 1 hot MTM plus a cold bag (with healthy snacks), with one day or more (depending on the 2 to 4x a week delivery schedule participant is on) also including 1 frozen MTM to total 5 meals per week.
  * Engagement: MOWCTX's trained volunteers and/or paid delivery drivers delivering the meals will have a brief social interaction ("check-in") with the participant.
  * MOWCTX Standard Wraparounds: Participants will have access to a case manager to assist with additional resources within the community and for additional support if needed (e.g., grocery shopping assistance, home repairs, and pet care).

SUMMARY:
This is a three-arm, parallel randomized trial study that will assess the impact of home delivery of medically-tailored meals (MTM) to community-dwelling older adults living with diabetes mellitus type 2 on measurements of diabetes control, mental health, and other exploratory outcomes such as healthcare use.

DETAILED DESCRIPTION:
This study aims to:

1. Assess the impact of medically-tailored meals program on diabetes management and mental health in comparison to usual care without such program.
2. Assess the differential impact of two delivery models being considered for payment by the health system on diabetes management and mental health: once-a-week frozen drop shipment model versus daily warm meal delivery model that is more complex to implement but allows for human connection and easier meal preparation.

Implementation of program:

Meals on Wheels (MoW) of Central Texas (MOWCTX) in Austin, Texas, will provide the meals and delivery service in this study. Meals are all medically tailored (diabetes friendly) and design by MOWCT's team of Registered Dietitians.

Participants:

Older adults, 55 and over, living in the Austin city limits with poorly controlled diabetes; Inclusion criteria:

* Adult 55-90
* Hemoglobin A1C >=7.5 (as measured at baseline)
* Living in Austin city limits and within a MOWCTX daily delivery route
* Interested and available to receive meals during delivery window time
* Has access to a freezer and a microwave
* Pass a MOWCTX background check

Trial:

Eligible participants will be recruited from selected Federally Qualified Health Centers in the Austin area, MOWCTX clients on waitlist, and other (e.g. Medicaid recipients).

Participants will be randomized to one of three arms: 1) Waitlisted control; 2) Weekly frozen drop shipment of MTM 3) Daily Warm delivery of MTM with in-person check-ins during delivery.

Phase 1 (first 6 months) The intervention arms will receive their assigned method of meal delivery (weekly frozen or daily warm), for a total of 10 meals a week, including two main meals per day and snacks. The control arm will not receive any meals during this phase. All arms will receive printed educational materials at baseline.

Phase 2 (month 6 to 12) All arms will receive 2-4 meals a week (depending on participant's availability) delivered via the traditional meal services from MOWCTX, which includes one hot meal plus a snack delivered daily. Meal delivery can also include 1 or more frozen meals to account for a total of 5 meals per week.

Primary outcome is Hemoglobin A1C and secondary outcomes include depression as measured by PHQ-8 and other mental health measures.

ELIGIBILITY:
Inclusion Criteria:

* Adult 55-90
* Hemoglobin A1c ≥7.5%
* Living in Austin city limits and within a MOWCTX daily delivery route
* Interested and available to receive meals during delivery window time
* Has access to a freezer and a microwave
* Pass a MOWCTX background check

Exclusion Criteria:

* Participated in MOW program in previous 3 months.
* Has any of the following: dementia or cognitive impairment, diagnosis of heart failure, cirrhosis, or active cancer
* Is receiving hospice care
* Does not pass a MOWCTX background check

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C (HbA1c) | Baseline to 6 months
  Finger stick point-of-care portable device.

SECONDARY OUTCOMES:
Change in Hemoglobin A1C | Baseline to 9 &12 months, 6 months to 12 months.
  Finger stick point-of-care portable device.
Program meal consumption | 6 months, 12 months
  For frozen and warm meals, self-report on what was actually consumed (customized survey)
Diet quality as assessed by NHANES DSQ | 6 months, 12 months
  Self-report of food consumption patterns
Loneliness as assessed by scores on the 3-item UCLA Loneliness Scale | 6 months, 12 months
  Respondents rate each item as 'Never' , 'Rarely', 'Sometimes' or 'Often'. Scores range from 3 to 9. Higher numbers imply greater loneliness.
Depressive symptoms as assessed by scores on the the 8-item Depression Health Questionnaire (PHQ-8) | 6 months, 12 months
  Respondents answer to eight questions that reflect the DSM-IV diagnosis criteria of depressive disorders. These questions ask how often in the past 2 weeks the respondent had experienced a particular depressive symptom. Each answer is scored from 0 to 3 and then summed. Total scores go from 0 and 24 points, with higher scores indicating greater depressive symptoms.
Anxiety symptoms as assessed by the 7-item Generalized Anxiety Disorder Scale (GAD-7) | 6 months
  Investigators will use the Generalized Anxiety Disorder Scale (GAD-7) to measure anxiety. Scored from 0-3, and a score of 0 indicates lower levels of anxiety while a score of 3 indicates higher levels of anxiety.
Diabetes Self-Efficacy as assessed by scores on the Stanford Self-Efficacy for Diabetes Scale 8-item | 6 months, 12 months
  Respondents are asked to score their level of confidence (scale from 1, not at all confident, to 10, totally confident) at the present time in doing tasks related to diabetes management (e.g., diet behavior, physical activity, measuring blood glycemia and others). Higher scores indicate higher self-efficacy.
Food security status as assessed by the USDA Food Security Survey Module: Six-Item Short Form | 6 months, 12 months
  Self-reported with a 30-day lookback period. The sum of affirmative responses to the six questions in the module is the household's raw score on the scale. Higher scores indicate greater food insecurity.
Health Status and Quality of Life as assessed by scores on Short-form 12-item (SF-12) | 6 months, 12 months
  Measures physical and mental health status. Summary scores range from 0-100, with higher scores indicating a better self-reported level of health.
Healthcare delay due to cost | 6 months, 12 months
  Self-report of delaying healthcare due to cost. 1 item.
Emergency room visits | 6 months, 12 months
  Self-report of going to a hospital emergency room.
Food-basic needs trade-offs (3 items) | 6 months, 12 months
  Self-report of trading off paying for food vs. paying for medicine or medical care, for utilities, and for housing
Medication underuse due to cost (2 items) | 6 months, 12 months
  Self-report of not acquiring a prescribed medication or took reduce dosage due to cost.

CONTACTS AND LOCATIONS:
Overall Officials: Maninder K Kahlon, PhD, Principal Investigator — University of Texas at Austin
Locations (2):
- United States (2):
  - Meals on Wheels Central Texas, Austin, Texas
  - CommUnityCare Health Centers (all Austin clinics), Austin, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04277117/Prot_SAP_001.pdf